CLINICAL TRIAL: NCT05062070
Title: A Phase I/II, Closed Label, Randomized, Pilot Study for the Safety and Efficacy of TolaSure Gel, 5% w/w Targeting Aggregated Mutant Keratin in Severe Epidermolysis Bullosa Simplex (TAMES)
Brief Title: Safety and Efficacy of Topical TolaSure Targeting Aggregated Mutant Keratin in Severe Epidermolysis Bullosa Simplex
Acronym: TAMES
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioMendics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TAMES-01
Record Dates: First submitted 2021-09-21; First posted 2021-09-30 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Epidermolysis Bullosa Simplex
Keywords: Epidermolysis Bullosa; Epidermolysis Bullosa Simplex; EBS; Severe EBS; EBS Dowling-Meara; Skin Diseases; Suction Blister; Skin Abnormalities; Keratin; Aggregate; Mutant; EBS-DM
MeSH Terms: conditions — Epidermolysis Bullosa Simplex; Epidermolysis Bullosa; Skin Diseases; Skin Abnormalities

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 5 Percent TolaSure Topical Gel (Active Comparator): 5% (w/w) TolaSure Gel
  Interventions: Drug: TolaSure Topical Gel
- Topical Vehicle Gel (Placebo Comparator): TolaSure Vehicle Gel
  Interventions: Drug: Vehicle Topical Gel

INTERVENTIONS:
Drug: TolaSure Topical Gel — TolaSure Topical Gel is applied once-daily for up to 10 weeks to designated Treatment Area and Suction Blister Area.
  Other Names: Active Ingredient BM-3103
  Arms: 5 Percent TolaSure Topical Gel
Drug: Vehicle Topical Gel — TolaSure Vehicle Gel is applied once-daily for up to 10 weeks to designated Treatment Area and Suction Blister Area.
  Other Names: TolaSure Vehicle Gel
  Arms: Topical Vehicle Gel

SUMMARY:
TolaSure is a topical gel for the promotion of accelerated wound healing. This Phase I study will assess the safety, tolerability, and clinical effects of TolaSure when applied to wounded skin areas of patients diagnosed with severe epidermolysis bullosa simplex (i.e., EBS-Dowling Meara). A total of 10, severe EBS patients, males and females ages 18 years and older, will be enrolled. Patients will apply TolaSure and Vehicle Gel once-daily for a maximum of 10 weeks.

DETAILED DESCRIPTION:
This is a closed-label, randomized, double-blind, Phase I clinical study to assess the safety and tolerability of the investigational product (IP), TolaSure Gel, 5% w/w, in patients diagnosed with severe epidermolysis bullosa simplex (EBS, previously known as EBS-Dowling Meara). Each patient (5 to complete) will apply TolaSure Gel, 5% w/w and TolaSure Vehicle Gel once-daily to defined Treatment Areas and Suction Blister Areas. End of Study (EOS) will occur at the Principal Investigator's (PI's) discretion according to the resolution or lack of improvement of the Treatment Areas. The maximum time a patient could be in the study is 10 weeks. The average time frame for each patient to complete the study is expected to be 6-8 weeks.

The primary safety endpoint will be the incidence of treatment-emergent adverse events (TEAEs). Safety monitoring will include physical exams, vital sign measurements, clinical laboratory testing (blood and urinalysis), and urine pregnancy testing (as appropriate).

Secondary efficacy endpoints will (1) assess wound severity within the Treatment Areas using an Investigator Global Assessment (IGA) scoring system, (2) examine under a microscope keratinocyte morphology and the incidence of keratin aggregates in Treatment Area skin biopsies, (3) determine the time required to induce a suction blister within the designated Suction Blister Areas, and (4) evaluate patient self-assessment of overall impression, pain, and itch within the Treatment Areas. The information obtained from these assessments will be used to examine the efficacy of TolaSure treatment in improving EBS symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Patient is a male or female at least 18 years of age.
* Patient has a documented genetic mutation in either the keratin 14 (K14) or keratin 5 (K5) gene and that their EBS diagnosis and/or specific mutation are consistent with severe EBS (previously EBS-DM). (If severe EBS is suspected but not genetically confirmed, confirmatory testing will be performed).
* Patient possesses the four required skin areas:

  * Treatment Areas:

    * Must have two (2) Treatment Areas defined as an IGA score ≥ 3. Treatment Areas may have defined erosions, erythema, and ulcerations.
    * Must be comparable in size with an area of approximately 300-400 cm^2 per area. Individually, a treatment area may be continuous or non-contiguous and must contain newly-formed blisters/erosions. Ideally, the two Treatment Areas on the patient should not be adjacent to each other and should be located bilaterally and roughly symmetrically on the trunk, abdomen, or upper or lower extremities.
    * May not be infected (as assessed by the Principal Investigator) or have been treated with a topical antibiotic within 14 days.
    * May not be located on palms, soles, scalp, groin, and any other areas that the Principal Investigator believes there will be difficulty in applying treatments and bandaging or assessing outcome measures.
  * Suction Blister Areas (SBAs):

    * Must have two (2) areas of non-wounded and visually uninvolved skin, defined as an IGA score of zero (0).
    * Must be comparable in size (approximately 50 cm^2)
* If the patient is a woman of childbearing potential (WOCBP),

  * Has a negative urine pregnancy test.
  * Agrees to use an approved effective form of birth control with failure rates <1% per year (e.g., implant, injectable, combined oral contraceptive, intrauterine contraceptive device, sexual abstinence, vasectomized partner) during participation in the study (and at least 3 months thereafter).
  * Is not nursing.
* Patient's laboratory values (blood and urine) are within the range of normal or abnormal values are within normal levels for the disease and in the opinion of the Principal Investigator the values are not clinically relevant for study participation.
* Patient is in good general health and free of any known disease state or physical condition which, in the Investigator's opinion, might impair evaluation of the EBS wounds or which exposes the patient to an unacceptable risk by study participation.
* Over the duration of the study, the patient agrees to not use any other topical therapies and/or impregnated dressings within the Treatment Areas or Suction Blister Areas (e.g., medicated cleansers, CBD oil, MediHoney, Silvadine cream 1%, topicals containing antimicrobials, keratin, and/or collagen, lipido-colloid or polymeric membrane dressings, and/or hydrogels).
* Patient must be able and willing to follow study procedures and instructions in order to maintain compliance throughout the study period.
* Patient has been informed, has read and understood the subject informed consent form, and has given written informed consent.

Exclusion Criteria:

* Patient's use of prior or concomitant medication or medical treatments/procedures:

  * Any investigational drug within 30 days.
  * Systemic steroidal therapy within 30 days.
  * Topical steroidal therapy within 14 days (Note: inhaled and ophthalmic products containing steroids are allowed).
  * Systemic antibiotic therapy within 7 days.
  * Systemic diuretics or cardiac glycosides within 30 days.
  * Currently receiving chemotherapy or radiation.
  * Patient has undergone stem cell transplant or gene therapy for the treatment of inherited EB.
  * Surgery within the previous 3 months (except for minor cosmetic or dental procedures).
* Patient's medical history includes:

  * Cancer that is currently undergoing treatment.
  * History of severe vitamin, mineral, or protein deficiency.
  * Current systemic infection.
  * HIV/AIDS.
  * Non-EBS skin disease (e.g., psoriasis, atopic dermatitis, eczema, sun damage, etc.), or condition (e.g., sunburn) that, in the opinion of the Investigator, might put the subject at undue risk by study participation or interferes with the study medication application or the study assessments.
  * An illness (e.g., neurological, cardiovascular, respiratory, hepatic, renal, or metabolic disease), condition, or situation that in the opinion of the Investigator is likely to interfere with the patient's participation in or completion of the study.
* Factors present in the patient and/or his/her legal representative that could interfere with study compliance such as inability to attend scheduled study visits or to perform study protocol procedures.
* Patient is a member of the investigational team or his/her immediate family.
* History of drug or alcohol abuse (as defined by the Investigator).
* Patient's use of smoking/vaping tobacco products.
* Other unspecified reasons that, in the opinion of the Investigator, make the subject unsuitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-06-22 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (TEAEs) | Day 1, Day 2, then Weekly until End of Study (maximum 10 weeks)
  Safety monitoring will include clinical chemistry tests, physical examinations (including assessment of Treatment and Suction Blister Areas), and vital sign measurements. These assessments along with AE reviews will identify potential TEAEs.

SECONDARY OUTCOMES:
Investigator Global Assessment (IGA) | Day 1, Day 2, then Weekly until End of Study (maximum 10 weeks)
  The Principal Investigator will use the IGA scale to score the average overall severity of the EBS wounds within the Treatment Areas, considered together. Changes from baseline in IGA scores for the TolaSure-treated and Vehicle-treated Treatment Areas will be analyzed.
Keratin Aggregate Counts and Cell Morphology Assessment | Day 1, During Study (optional, estimated Week 3-Week 6), End of Study (maximum 10 weeks)
  Biopsies from perilesional skin in each of the Treatment Areas are examined to determine a change from baseline in the number of keratin aggregate positive basal and suprabasal keratinocytes using transmission electron microscopy (TEM) and/or light microscopy.
Suction Blister Time | Day 1 and End of Study (maximum 10 weeks)
  A suction blister is raised within the Suction Blister Areas and the time to blister formation is recorded in seconds. Changes from baseline suction blister times in the TolaSure-treated and Vehicle-treated Suction Blister Areas will be analyzed.
Patient's-reported Overall Impression Score of Treatment Areas | Day 1, then Weekly until End of Study (maximum 10 weeks)
  Change from baseline in the patient-reported overall impression score of both the TolaSure-treated and Vehicle-treated Treatment Areas will be calculated.
Patient's-reported Pain Score of Treatment Areas | Day 1, then Weekly until End of Study (maximum 10 weeks)
  Change from baseline in the patient-reported pain numerical rating scale (NRS) of both the TolaSure-treated and Vehicle-treated Treatment Areas will be calculated.
Patient's-reported Itch Score of Treatment Areas | Day 1, then Weekly until End of Study (maximum 10 weeks)
  Change from baseline in the patient-reported itch numerical rating scale (NRS) of both the TolaSure-treated and Vehicle-treated Treatment Areas will be calculated.

OTHER OUTCOMES:
Proportion of Keratinocytes containing Autophagosomes | Day 1, During Study (optional, estimated Week 3-Week 6), End of Study (maximum 10 weeks)
  Biopsies from perilesional skin in each of the Treatment Areas are examined to determine a change from baseline in the number of autophagosome positive basal and suprabasal keratinocytes using transmission electron microscopy (TEM) and/or light microscopy.
Cytokine Content in Suction Blister Fluid | Day 1 and End of Study (maximum 10 weeks)
  Suction blister fluid collected from each of the induced suction blisters will be used to determine a change from baseline in inflammatory cytokine content.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University School of Medicine, Dermatology Department, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No